CLINICAL TRIAL: NCT04173078
Title: Computerized Intervention for Distress Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Florida State University (Other)
Responsible Party: Principal Investigator, Richard Macatee, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201720828; F31DA039644-01A1 (NIH)
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Cannabis Use Disorder
Keywords: distress intolerance; stress

STUDY DESIGN:
Intervention Model Description: At the end of the baseline assessment, the participant was randomized to the Computerized Distress Intolerance Intervention condition or the Computerized Healthy Behaviors condition. Participants in each condition attended two 1-hour intervention sessions followed by a post-treatment assessment. Follow-up assessments were conducted one-month and four-months after the post-treatment assessment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blind to whether they were in the experimental (Distress Intolerance Intervention) or control (Healthy Behaviors Intervention) condition. All outcome measures were self-report except for the four-month follow-up Cannabis Use Diagnostic interview which was conducted by an interviewer blind to the participant's treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Distress Intolerance Intervention (Experimental): Two, 1-hour computerized sessions that include psychoeducation about emotional avoidance, idiographic emotional exposure, and construction of idiographic implementation intentions to practice distress tolerance skills outside of session.
  Interventions: Behavioral: Computerized Distress Intolerance Intervention
- Computerized Healthy Behaviors Intervention (Placebo Comparator): Two, 1-hour computerized sessions that focus on psychoeducation about the importance of a healthy lifestyle.
  Interventions: Behavioral: Computerized Healthy Behaviors Intervention

INTERVENTIONS:
Behavioral: Computerized Distress Intolerance Intervention
  Arms: Computerized Distress Intolerance Intervention
Behavioral: Computerized Healthy Behaviors Intervention
  Arms: Computerized Healthy Behaviors Intervention

SUMMARY:
This study evaluates the impact of a computerized distress intolerance intervention relative to a control intervention on cannabis use-related behavior and neurophysiology.

DETAILED DESCRIPTION:
Distress intolerant cannabis users were randomized to a computerized distress intolerance intervention or a control intervention. Primary and secondary outcomes consist of the treatment target, cannabis use-related behavior, and theoretically-relevant neurophysiological processes (i.e., cannabis cue reactivity, response inhibition).

ELIGIBILITY:
Inclusion Criteria:

* Distress Intolerance Index score >= 20
* Average cannabis use frequency in the past year >= 2-3/week

Exclusion Criteria:

* Current suicidal ideation
* History of psychotic symptoms
* Bipolar-spectrum disorder without stabilization on medication for >= 3 months
* Change in psychotropic medication in the past month
* Current CBT for internalizing or substance use disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Distress Intolerance Index (DII) score from Baseline through 4-Month Follow-Up | Baseline, post-treatment (i.e., ~1 week following the last treatment session), 1-month follow-up, 4-month follow-up
  Self-report measure of Distress Intolerance (Distress Intolerance Index [DII]; McHugh & Otto, 2012). The DII is a self-report measure comprised of 10 items that are summed together to form a total score (minimum: 0; maximum: 40). Higher scores indicate greater distress intolerance (i.e., worse outcome).
Change in Mirror-Tracing Persistence Task (MTPT) quit latency from Baseline to Post-Treatment | Baseline, post-treatment (i.e., ~1 week following the last treatment session)
  Behavioral measure of Distress Intolerance (Mirror-Tracing Persistence Task [MTPT]; Macatee & Cougle, 2015). The MTPT is a behavioral persistence measure that assesses behavioral distress intolerance via the latency to quit a distressing task. Scores range from 0 seconds to a maximum persistence time of 7 minutes. Lower scores indicate greater distress intolerance (i.e., worse outcome).
Change in Marijuana Problems Scale (MPS) score from Baseline through 4-Month Follow-Up | Baseline, post-treatment (i.e., ~1 week following the last treatment session), 1-month follow-up, 4-month follow-up
  Self-report measure of marijuana use-related problems (Marijuana Problems Scale [MPS]; Stephens et al., 2000). The MPS is a self-report measure of marijuana use-related problem severity in the past month. The measure is comprised of 19 items with a minimum score of 0 and a maximum score of 38. Higher scores indicate greater marijuana use-related problem severity in the past month (i.e., worse outcome).
Change in Cannabis Use Disorder (CUD) diagnostic criteria from Baseline to 4-Month Follow-Up | Baseline, 4-month follow-up
  Interviewer-assessed Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Cannabis Use Disorder diagnostic criteria. DSM-5 Cannabis Use Disorder criteria were assessed via interview at baseline and again at the 4-month follow-up. Total number of Cannabis Use Disorder criteria was used to assess Cannabis Use Disorder severity (minimum score: 0; maximum score: 11). Higher scores indicate greater Cannabis Use Disorder severity (i.e., worse outcome).
Change in Timeline follow-back (TLFB) cannabis use frequency from Baseline through 4-Month Follow-Up | Baseline, post-treatment (i.e., ~1 week following the last treatment session), 1-month follow-up, 4-month follow-up
  Percent cannabis use days in the past month (Timeline follow-back [TLFB]; Hjorthoj et al., 2012). The Timeline follow-back (TLFB) is a self-report measure that assesses cannabis use over the past 4 weeks. Percentage of days on which cannabis was used in the past four weeks was used to assess cannabis use frequency (minimum: 0%; maximum: 100%). Higher scores indicate greater cannabis use frequency (i.e., worse outcome).
Change in Marijuana Motives Measure (MMM) score from Baseline through 4-Month Follow-Up | Baseline, post-treatment (i.e., ~1 week following the last treatment session), 1-month follow-up, 4-month follow-up
  Self-reported motives for cannabis use (Marijuana Motives Measure [MMM]; Zvolensky et al., 2007). The Marijuana Motives Measure (MMM) is a self-report measure that assesses different motives for marijuana use. The coping motives subscale was the subscale of interest in this project. The Coping motives subscale is comprised of 4 items that are then averaged (minimum score: 1; maximum score: 5). Greater scores indicate greater coping motives for marijuana use (i.e., worse outcome).
Change in Marijuana Craving Questionnaire (MCQ) score from Baseline to Post-Treatment | Baseline, post-treatment (i.e., ~1 week following the last treatment session)
  Self-reported state craving for marijuana (Marijuana Craving Questionnaire [MCQ]; Heishman et al., 2009). The Marijuana Craving Questionnaire (MCQ) is a self-report measure of current craving for marijuana use. The emotionality subscale was the subscale of interest in this project. The Emotionality subscale is comprised of 5 items that are then averaged (minimum score: 1; maximum score: 7). Greater scores indicate greater marijuana craving (i.e., worse outcome). In this project, the outcome of interest is the extent to which a laboratory stress induction increases state marijuana craving.

SECONDARY OUTCOMES:
Change in electroencephalography (EEG) index of acute stress modulation of cannabis cue reactivity (assessed by the Late Positive Potential [LPP]) from Baseline to Post-Treatment | Baseline, post-treatment (i.e., ~1 week following the last treatment session)
  Acute Stress modulation of the Late Positive Potential (LPP) to Cannabis Cues. The LPP to visual cannabis cues before and after a laboratory stress induction will be measured as a neurophysiological index of acute stress modulation of cannabis cue incentive salience. Greater values indicate a larger neural response to cannabis cues during acute stress (i.e., worse outcome).
Change in electroencephalography (EEG) index of acute stress modulation of threat reactivity (assessed by the Late Positive Potential [LPP]) from Baseline to Post-Treatment | Baseline, post-treatment (i.e., ~1 week following the last treatment session)
  Acute Stress modulation of the Late Positive Potential (LPP) to threat stimuli. The LPP to visual threat stimuli before and after a laboratory stress induction will be measured as a neurophysiological index of acute stress modulation of threat reactivity. Greater values indicate a larger neural response to threat during acute stress (i.e., worse outcome).
Change in electroencephalography (EEG) index of acute stress modulation of response inhibition (assessed by the N200 [N2]) from Baseline to Post-Treatment | Baseline, post-treatment (i.e., ~1 week following the last treatment session)
  Acute stress modulation of the N2 to no-go stimuli. The N2 to no-go vs. go stimuli on a go/no-go task before and after a laboratory stress induction will be measured as a neurophysiological index of the acute stress modulation of response inhibition. More negative values indicate a larger neural response to stimuli requiring response inhibition during acute stress (i.e., better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Macatee, PhD, Principal Investigator — Auburn University

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be made available upon request once primary and secondary outcome manuscripts have been published.

REFERENCES:
- [Background] McHugh RK, Otto MW. Refining the measurement of distress intolerance. Behav Ther. 2012 Sep;43(3):641-51. doi: 10.1016/j.beth.2011.12.001. Epub 2011 Dec 20. PMID 22697451
- [Background] Macatee RJ, Cougle JR. Development and evaluation of a computerized intervention for low distress tolerance and its effect on performance on a neutralization task. J Behav Ther Exp Psychiatry. 2015 Sep;48:33-9. doi: 10.1016/j.jbtep.2015.01.007. Epub 2015 Jan 26. PMID 25681579
- [Background] Stephens RS, Roffman RA, Curtin L. Comparison of extended versus brief treatments for marijuana use. J Consult Clin Psychol. 2000 Oct;68(5):898-908. PMID 11068976
- [Background] Hjorthoj CR, Hjorthoj AR, Nordentoft M. Validity of Timeline Follow-Back for self-reported use of cannabis and other illicit substances--systematic review and meta-analysis. Addict Behav. 2012 Mar;37(3):225-33. doi: 10.1016/j.addbeh.2011.11.025. Epub 2011 Nov 26. PMID 22143002
- [Background] Zvolensky MJ, Vujanovic AA, Bernstein A, Bonn-Miller MO, Marshall EC, Leyro TM. Marijuana use motives: A confirmatory test and evaluation among young adult marijuana users. Addict Behav. 2007 Dec;32(12):3122-30. doi: 10.1016/j.addbeh.2007.06.010. Epub 2007 Jun 9. PMID 17602842
- [Background] Heishman SJ, Evans RJ, Singleton EG, Levin KH, Copersino ML, Gorelick DA. Reliability and validity of a short form of the Marijuana Craving Questionnaire. Drug Alcohol Depend. 2009 Jun 1;102(1-3):35-40. doi: 10.1016/j.drugalcdep.2008.12.010. Epub 2009 Feb 13. PMID 19217724
- [Derived] Macatee RJ, Preston TJ, Afshar K, Schmidt NB, Cougle JR. Impact of a computerized distress intolerance intervention on electrocortical reactivity to cannabis and threat cues: A randomized controlled trial. Psychol Addict Behav. 2022 Nov;36(7):920-929. doi: 10.1037/adb0000815. Epub 2022 Feb 7. PMID 35129994